CLINICAL TRIAL: NCT05687643
Title: Shear Load In-shoe Plantar Sensing/Strain Analyses and Mapping in Diabetic Foot Ulcers
Acronym: SLIPSTREAM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: VS21/143856
Record Dates: First submitted 2022-09-28; First posted 2023-01-18 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Diabetic Foot; Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic Foot Ulcer (DFU) group: Inclusion criteria:
  1. Age >18
  2. A diagnosis of diabetes mellitus
  3. A diagnosis of diabetic peripheral neuropathy
  4. Recently healed plantar ulcer (within the last 3 months)
- Low risk group: Inclusion criteria:
  1. Age >18
  2. A diagnosis of diabetes mellitus
  3. Low risk for DFU according to the NG19 guidelines (no risk factors for ulceration except callus alone)

SUMMARY:
Stain Analysis Mapping of the Plantar surface (STAMP) is a method designed by the University of Leeds to measure 'in-shoe' strain patterns on the plantar surface of the foot. Shear Load Inductive Plantar Sensing (SLIPS) is an insole designed by the University of Leeds to measure plantar shear stress and plantar pressure. This study aims to compare plantar strain using STAMP and plantar shear stress and plantar pressure using SLIPS in two groups of patients with diabetes; high risk patients with a recently healed plantar ulcer and low risk patients (according to the NICE definition).

DETAILED DESCRIPTION:
Stain Analysis Mapping of the Plantar surface (STAMP) is a method designed by the University of Leeds to measure 'in-shoe' strain patterns on the plantar surface of the foot. The insole comprises a pseudorandom pattern applied to a plastically deformable insole using a temporary tattoo layer. STAMP utilises digital image correlation to track the deformation of the pattern following a period of walking.

Shear Load Inductive Plantar Sensing (SLIPS) is an insole designed by the University of Leeds to measure plantar shear stress and plantar pressure. SLIPS is an insole which integrates 64 tri-axis soft force sensors which simultaneously measures shear stress and pressure. The SLIPS insole has been designed to measure the plantar load of the right foot and due to its size can only be accommodated by a size 8-11 shoe.

The commercial device Pedar (Novel gmbh) will be used as a reference for plantar pressure measurement in both groups.

This study aims to compare plantar strain using STAMP and plantar shear stress and plantar pressure using SLIPS in two groups of patients with diabetes; high risk patients with a recently healed plantar ulcer and low risk patients (according to the NICE definition).

It is hypothesised that patients with a recently healed plantar ulcer with exhibit elevated plantar strain, plantar shear stress and plantar pressure than the low risk group.

ELIGIBILITY:
DFU group:

Patients will undergo STAMP and Pedar assessment if they fulfil the following criteria.

Inclusion Criteria:

1. Age >18
2. A diagnosis of diabetes mellitus
3. A diagnosis of diabetic peripheral neuropathy
4. Recently healed plantar ulcer (within the last 3 months)
5. Able to provide informed consent
6. Previous open or endovascular revascularisation

SLIPS inclusion criteria:

Patients will also undergo assessment with the SLIPS insole if they fulfil the following inclusion criteria:

1. Recently healed plantar DFU located on the right foot
2. The right foot can be accommodated in a size 8-11 shoe
3. Weight <100kg

Low risk group:

Patients will undergo STAMP and Pedar assessment if they fulfil the following criteria:

1. Age >18
2. A diagnosis of diabetes mellitus
3. Low risk for DFU according to the NICE NG 19 guidelines (no risk factors for ulceration except callus alone)
4. Able to provide informed consent

Exclusion Criteria:

1. Unable to mobilise independently 150m without the use of walking aids and thus unable to complete the walking assessments
2. Previous ipsilateral minor amputation
3. Previous ipsilateral surgical offloading procedure
4. Previous contralateral major amputation
5. Ipsilateral toe pressure <40mmHg

SLIPS assessment inclusion:

1. The right foot can be accommodated in a size 8-11 shoe
2. Weight <100kg

Exclusion criteria:

1. Unable to mobilise independently 150m without the use of walking aids and thus unable to complete the walking assessments
2. Previous ipsilateral minor amputation
3. Presence of a foot deformity
4. Previous contralateral major amputation
5. Ipsilateral toe pressure <40mmHg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: DFU group:
  Patients with a recently healed plantar ulcer recruited from a specialised Diabetes Limb Salvage Service in a tertiary referral centre.
  Low risk group:
  Patients with diabetes and low risk for ulceration recruited from the community podiatry service.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-04-03 (Estimated); Study Completion 2024-04-03 (Estimated)

PRIMARY OUTCOMES:
Peak plantar strain | At clinical visit on study entry
  The difference in peak plantar strain (%) (as measured with STAMP) between the DFU and low risk group

SECONDARY OUTCOMES:
Regional peak plantar strain | At clinical visit on study entry
  The difference in regional peak plantar strain (%) between the DFU and low risk group at the 10 pre-specified regions: heel, midfoot, 1st metatarsal head (MTH), 2nd MTH, 3rd MTH, 4th MTH, 5th MTH, hallux, 2nd toe, toes 3-5
Regional peak plantar shear | At clinical visit on study entry
  The difference in regional peak plantar shear (kPa) between the DFU and low risk group at the 10 pre-specified regions: heel, midfoot, 1st metatarsal head (MTH), 2nd MTH, 3rd MTH, 4th MTH, 5th MTH, hallux, 2nd toe, toes 3-5
Peak Plantar pressure | At clinical visit on study entry
  Global peak plantar pressure (kPa) between DFU and low risk groups.
Regional Peak Plantar pressure | At clinical visit on study entry
  Regional peak plantar pressure (kPa) between DFU and low risk groups

CONTACTS AND LOCATIONS:
Overall Officials: David A Russell, Principal Investigator — University of Leeds
Locations (1):
- Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/43/NCT05687643/Prot_SAP_000.pdf